CLINICAL TRIAL: NCT00108537
Title: Non-Nicotine Agents for Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ADRD-013-01S
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2006-10

CONDITIONS: Tobacco Use Disorder
Keywords: smoking; nicotine; drug therapy; smoking cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation | interventions — Bupropion; Transdermal Patch; Nicotine

INTERVENTIONS:
Drug: bupropion and transdermal patch
Drug: transdermal patch and nicotine inhaler

SUMMARY:
The primary objective of this study is to determine which is the better approach to smoking cessation in veterans: bupropion combined with transdermal nicotine or high dose nicotine replacement therapy (NRT) using transdermal nicotine combined with nicotine inhaler.

DETAILED DESCRIPTION:
This study is a two-arm open-label, randomized controlled trial of bupropion combined with transdermal nicotine versus high dose NRT (transdermal nicotine and nicotine inhaler) with all subjects receiving a behavioral counseling program for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Readiness to set a quit date in the next two weeks,
* Current smoking of at least 15 cigarettes a day

Exclusion Criteria:

* Current untreated depression or receiving treatment for depression,
* History of seizures, major head injury, or other predisposition for seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- Denver VA Medical Center, Denver, Colorado, United States